CLINICAL TRIAL: NCT03704428
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, MAD Study to Evaluation of Safety, Tolerability and PK of SHR1314 With Axial Spondyloarthritis
Brief Title: Safety, Tolerability and PK of SHR1314 in axSpA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1314-AS-102
Record Dates: First submitted 2018-09-24; First posted 2018-10-12 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2018-01

CONDITIONS: Axial Spondyloarthritis
Keywords: SHR1314
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Multiple subcutaneous injections of SHR-1314 dose 1
  Interventions: Drug: SHR-1314
- Cohort 2 (Experimental): Multiple subcutaneous injections of SHR-1314 dose 2
  Interventions: Drug: SHR-1314
- Cohort 3 (Experimental): Multiple subcutaneous injections of SHR-1314 dose 3
  Interventions: Drug: SHR-1314
- Cohort 4 (Experimental): Multiple subcutaneous injections of SHR-1314 dose 4
  Interventions: Drug: SHR-1314
- Cohort 5 (Experimental): Multiple subcutaneous injections of SHR-1314 dose 5
  Interventions: Drug: SHR-1314

INTERVENTIONS:
Drug: SHR-1314 — Pharmaceutical form: Injection solution. Route of administration: subcutaneous injection.
  Other Names: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety, Tolerability and Pharmacokinetics (PK) of SHR1314 with axial spondyloarthritis.

DETAILED DESCRIPTION:
This was a phase I, multicenter, double-blind, randomized, placebo-controlled study. The study originally planned to enroll 5 cohorts of 8 subjects each (N=40).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of axial spondyloarthritis (axSpA) and fulfilling the 2009 ASAS classification criteria.
2. Have a history of back pain ≥3 months with age at onset <45 years.
3. Have active axSpA defined as BASDAI ≥4 at screening and baseline.
4. Have objective signs of inflammation by presence of elevated ESR and/or presence of elevated CRP.
5. In the past had an inadequate response to at least 1 or 2 non-steroidal anti-inflammatory drugs (NSAIDS) for duration of 4 weeks or cannot tolerate NSAIDS.
6. If taking NSAIDS be on stable dose for at least 2 weeks prior to randomization.

Exclusion Criteria:

1. History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection.
2. Previous exposure to other biologic drug directly targeting Interleukin (IL)-17 or Interleukin (IL)-17 receptor.
3. Total ankylosis of the spine.
4. Have recently received biologics, tumor necrosis factor inhibitors or other immunomodulatory agents within 12 weeks.
5. Have either a current diagnosis or a recent history of malignant disease.
6. Are pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of multiple subcutaneous injections of SHR1314 in adult patients with axial spondyloarthritis 1.Incidence of Treatment-Emergent Adverse Events 2.Incidence of Injection site reaction | Baseline to 169 days after dose administration
  Safety and tolerability of multiple subcutaneous injections of SHR1314 assessed by adverse events and serious adverse events.
  1. Incidence of Treatment-Emergent Adverse Events
  2. Incidence of Injection site reaction

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of SHR-1314 | Baseline to 169 days after dose administration
  maximum concentration (Cmax)
Time to maximum observed serum concentration (tmax) of SHR-1314 | Baseline to 169 days after dose administration
  Time to maximum concentration (Tmax)
Time to elimination half-life (t1/2) of SHR-1314 | Baseline to 169 days after dose administration
  t1/2
Assessment of development of Anti-drug Antibodies (ADAs) | Baseline to 169 days after dose administration
  Incidence of development of Anti-drug Antibodies (ADAs)
Proportion of Participants Achieving an ASAS20 Response | Week2, 4, 6, 8, 12,16
  ASAS20 Response

CONTACTS AND LOCATIONS:
Overall Officials: Fei Sun, MD, Principal Investigator — People's Liberation Army General Hospital; Xin Chang, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- Jianwen Chen, Shanghai, China

IPD SHARING:
Plan to Share IPD: No